CLINICAL TRIAL: NCT04846114
Title: Efficacy of Local Hemostatic Management in Implant Surgery in Anticoagulated Patients on Warfarin: a Randomized Clinical Study
Brief Title: Dental Implants in Patients Under Oral Anticoagulant Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jorge Ernesto Aguilar (Other)
Responsible Party: Sponsor-Investigator, Jorge Ernesto Aguilar, Director and Professor, Oral Implantology Program, Universidad del Salvador, Argentina
Organization: Universidad del Salvador, Argentina (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VRID 1500
Record Dates: First submitted 2021-04-11; First posted 2021-04-15 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Oral Anticoagulant Therapy
Keywords: Dental Implants; Anticoagulant Therapy; Warfarin; Tranexamic Acid; Bismuth subgallate

STUDY DESIGN:
Intervention Model Description: 80 surgical procedures (pr) in 71 patients (18 not OAT/53 on OAT) were assigned to one of four groups: control group (Cg n=20 pr not OAT) and 3 experimental groups of patients on OAT with local hemostatic management were randomized: tranexamic acid group (TXAg n=20 pr), bismuth subgallate group (BSg n=20 pr) and dry gauze group (DGg n=20 pr).
Who Masked: Participant
Masking Description: The participants on OAT allocated to one of the three different local hemostatic strategies, were not informed wich agent was used. Time of compression was equal in all groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Cg) (Active Comparator): The control group (Cg) comprised 20 procedures performed in patients not on OAT.
  Buccal and palatal-lingual flaps were repositioned and sutured with simple stitches using 5/0 monofilament nylon yarn, and a dry gauze was applied for 30 minutes.
  Interventions: Procedure: Dental implant surgery
- Tranexamic acid group (TXAg) (Experimental): TXAg group comprised 20 procedures performed in patients OAT. Buccal and palatal-lingual flaps were repositioned and sutured as in the Cg plus compression on the wound for 30 minutes using a gauze soaked in the contents of a 500mg ampoule of TXA, after which a new gauze soaked in the contents of a 500mg ampoule of TXA was applied for two hours.
  Interventions: Procedure: Dental implant surgery
- Bismuth subgallate group (BSg) (Experimental): BSg group comprised 20 procedures performed in patients OAT. At the moment of surgery, the contents of an anestube (1.8 ml) were mixed with a sufficient amount of BS powder to obtain a paste similar in consistency to tooth-paste (29). A thin layer of the paste was applied on the bone ridge, and buccal and palatal-lingual flaps were then repositioned and sutured as in the Cg. compression on the wound with a dry gauze for 30 minutes, after which a new dry gauze was placed for another two hours.
  Interventions: Procedure: Dental implant surgery
- Dry gauze group (DGg) (Experimental): DGg group comprised 20 procedures performed in patients OAT. Buccal and palatal-lingual flaps were repositioned and sutured as in the Cg plus compression on the wound with a dry gauze for 30 minutes, after which a new dry gauze was placed for another two hours.
  Interventions: Procedure: Dental implant surgery

INTERVENTIONS:
Procedure: Dental implant surgery

SUMMARY:
This study evaluated the outcomes in the post-operative recovery following dental implant surgery in patients who continued on oral anticoagulated therapy (OAT) with warfarin. The primary outcome of this study was to evaluate bleeding within the first 5 days post-surgery and presence of intraoral/extraoral hematomas in skin and mucosa oral.

DETAILED DESCRIPTION:
The aim of this study was compare: 1) the frequency of immediate and short term postoperative bleeding using tranexamic acid (TXAg), bismuth subgallate (BSg) or dry gauze (DGg) as local hemostatic 2) explore the relation between bleeding and the occurrence of hematomas, with length of incision, duration of surgery, and alveolar ridge recontouring. 80 surgical procedures performed in a total of 71 patients (20 surgical procedures in 18 patients not on OAT and 60 surgical procedures performed in 53 patients on OAT) that were assigned to one of four groups, so that each group included 20 procedures. The control group (Cg) comprised 20 procedures performed in patients not on OAT. The 60 procedures to be performed in patients on OAT were randomly to one of the three following experimental groups: 1) TXAg group, OAT plus TXA as local hemostatic agent; 2) BSg group, OAT plus BS as local hemostatic agent; 3) DGg group, OAT plus compression with dry gauze as local hemostatic agent. Outcomes variables were:

Intraoperative variables: length of incision expressed (Li) alveolar ridge recontouring (Arr), total duration of surgery (Ds), surgical quadrant and implant location.

Postoperative variables: immediate postoperative bleeding (within the first 30 minutes after surgery), short-term bleeding: within the first 5 days post-surgery, determined according to the index described by Bacci, presence of intraoral/extraoral hematomas in skin or mucosa. Descriptive statistical, analysis of variance and regression logistic analysis was performed. Statistical significance was set at a value of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

Subjects:

* Systemically healthy.
* Healthy periodontal tissues or well-controlled periodontal health.
* In need of a maximum of two dental implants per hemiarcade,
* Showing ≥8mm bone height and ≥6 horizontal bone width.
* Needing a maximum of two surgical procedures.
* Who had written consent from the referring service to undergo the surgical procedure.

Exclusion Criteria:

Subjects:

* Requiring implant placement immediately after extraction.
* Systemic disease contraindicating implant surgery.
* Mental disability preventing them from complying with the protocol.
* Hematological, metabolic, autoimmune or bone diseases.
* Hepatic alterations or receiving medication affecting liver function.
* Receiving corticoid therapy, chemotherapy, or anticoagulant therapy within 10 days prior to the surgery.
* Taking antibiotics that interact with oral anticoagulants.
* Requiring vertical or periosteal incisions.
* Requiring bone regeneration strategy.

When treatment involved placing an implant in more than one hemiarcade, the corresponding surgeries were scheduled 30 days apart.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Number of immediate postoperative bleeding events | Within the first 30 minutes after surgery
  0: no bleeding; -1: mild bleeding defined as minor oozing from the wound incision controlled with compressive gauze only -2: moderate bleeding associated with the presence of large clots continuously disrupting the surgical area and requiring additional hemostatic measures; -3: severe bleeding requiring further medical control of coagulation
Number of short-term bleeding events | Within the first 5 days post-surgery
  0: no bleeding; -1: mild bleeding defined as minor oozing from the wound incision controlled with compressive gauze only -2: moderate bleeding associated with the presence of large clots continuously disrupting the surgical area and requiring additional hemostatic measures; -3: severe bleeding requiring further medical control of coagulation
Number of presence of intraoral hematomas events | On day 7 post-surgery
  changes in mucosa color and edema (recorded as a dichotomous variable- yes/no).
Number of presence of extraoral hematomas events | On day 7 post-surgery
  changes in skin color and edema (recorded as a dichotomous variable- yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Aguilar, Chair Prof, Study Director — Universidad del Salvador; Mariano Vassallo, Assoc Prof, Principal Investigator — Universidad del Salvador; Jose Zamberlin, Assoc Prof, Principal Investigator — Universidad del Salvador; Marina Diaz Roig, Assist Prof, Principal Investigator — Universidad del Salvador; Ricardo Macchi, Chair Prof, Study Chair — University of Buenos Aires
Locations (1):
- Masters in Dental Implantology (MIO) program at the University of Salvador (USAL)-Argentine Dental Association, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keeling D, Baglin T, Tait C, Watson H, Perry D, Baglin C, Kitchen S, Makris M; British Committee for Standards in Haematology. Guidelines on oral anticoagulation with warfarin - fourth edition. Br J Haematol. 2011 Aug;154(3):311-24. doi: 10.1111/j.1365-2141.2011.08753.x. Epub 2011 Jun 14. No abstract available. PMID 21671894
- [Result] van Diermen DE, van der Waal I, Hoogvliets MW, Ong FN, Hoogstraten J. Survey response of oral and maxillofacial surgeons on invasive procedures in patients using antithrombotic medication. Int J Oral Maxillofac Surg. 2013 Apr;42(4):502-7. doi: 10.1016/j.ijom.2012.09.018. Epub 2012 Nov 2. PMID 23123097
- [Result] Caliskan M, Tukel HC, Benlidayi ME, Deniz A. Is it necessary to alter anticoagulation therapy for tooth extraction in patients taking direct oral anticoagulants? Med Oral Patol Oral Cir Bucal. 2017 Nov 1;22(6):e767-e773. doi: 10.4317/medoral.21942. PMID 29053656
- [Result] Madrid C, Sanz M. What influence do anticoagulants have on oral implant therapy? A systematic review. Clin Oral Implants Res. 2009 Sep;20 Suppl 4:96-106. doi: 10.1111/j.1600-0501.2009.01770.x. PMID 19663955
- [Result] Mehra P, Cottrell DA, Bestgen SC, Booth DF. Management of heparin therapy in the high-risk, chronically anticoagulated, oral surgery patient: a review and a proposed nomogram. J Oral Maxillofac Surg. 2000 Feb;58(2):198-202. doi: 10.1016/s0278-2391(00)90339-2. PMID 10670599
- [Result] George C, Barras M, Coombes J, Winckel K. Unfractionated heparin dosing in obese patients. Int J Clin Pharm. 2020 Apr;42(2):462-473. doi: 10.1007/s11096-020-01004-5. Epub 2020 Mar 5. PMID 32140914
- [Result] Daniels PR. Peri-procedural management of patients taking oral anticoagulants. BMJ. 2015 Jul 14;351:h2391. doi: 10.1136/bmj.h2391. PMID 26174061
- [Result] Halpern LR, Adams DR, Clarkson E. Treatment of the Dental Patient with Bleeding Dyscrasias: Etiologies and Management Options for Surgical Success in Practice. Dent Clin North Am. 2020 Apr;64(2):411-434. doi: 10.1016/j.cden.2019.12.010. Epub 2020 Jan 31. PMID 32111278
- [Result] Dewan K, Bishop K, Muthukrishnan A. Management of patients on warfarin by general dental practitioners in South West Wales: continuing the audit cycle. Br Dent J. 2009 Feb 28;206(4):E8; discussion 214-5. doi: 10.1038/sj.bdj.2009.112. Epub 2009 Feb 13. PMID 19214196
- [Result] Suresh V, Bishawi M, Manning MW, Patel C, Rogers J, Milano C, Schroder J, Daneshmand M, Powers D. Management of Patients With Left Ventricular Assist Devices Requiring Teeth Extraction: Is Halting Anticoagulation Appropriate? J Oral Maxillofac Surg. 2018 Sep;76(9):1859-1863. doi: 10.1016/j.joms.2017.10.022. Epub 2017 Oct 31. PMID 29156176
- [Result] Kammerer PW, Frerich B, Liese J, Schiegnitz E, Al-Nawas B. Oral surgery during therapy with anticoagulants-a systematic review. Clin Oral Investig. 2015 Mar;19(2):171-80. doi: 10.1007/s00784-014-1366-3. Epub 2014 Nov 22. PMID 25413495
- [Result] Lopez MA, Andreasi Bassi M, Confalone L, Gaudio RM, Lombardo L, Lauritano D. Clinical outcome of 215 transmucosal implants with a conical connection: a retrospective study after 5-year follow-up. J Biol Regul Homeost Agents. 2016 Apr-Jun;30(2 Suppl 1):55-60. PMID 27469549
- [Result] Ascani A, Iorio A, Agnelli G. Withdrawal of warfarin after deep vein thrombosis: effects of a low fixed dose on rebound thrombin generation. Blood Coagul Fibrinolysis. 1999 Jul;10(5):291-5. PMID 10456621
- [Result] Doonquah L, Mitchell AD. Oral surgery for patients on anticoagulant therapy: current thoughts on patient management. Dent Clin North Am. 2012 Jan;56(1):25-41, vii. doi: 10.1016/j.cden.2011.06.002. PMID 22117941
- [Result] Garcia DA, Regan S, Henault LE, Upadhyay A, Baker J, Othman M, Hylek EM. Risk of thromboembolism with short-term interruption of warfarin therapy. Arch Intern Med. 2008 Jan 14;168(1):63-9. doi: 10.1001/archinternmed.2007.23. PMID 18195197
- [Result] Akopov SE, Suzuki S, Fredieu A, Kidwell CS, Saver JL, Cohen SN. Withdrawal of warfarin prior to a surgical procedure: time to follow the guidelines? Cerebrovasc Dis. 2005;19(5):337-42. doi: 10.1159/000085027. Epub 2005 Apr 8. PMID 15818034
- [Result] Wahl MJ. Dental surgery in anticoagulated patients. Arch Intern Med. 1998 Aug 10-24;158(15):1610-6. doi: 10.1001/archinte.158.15.1610. PMID 9701094
- [Result] Wahl MJ. Demystifying medical complexities. J Calif Dent Assoc. 2000 Jul;28(7):510-8. PMID 11324133
- [Result] Clemm R, Neukam FW, Rusche B, Bauersachs A, Musazada S, Schmitt CM. Management of anticoagulated patients in implant therapy: a clinical comparative study. Clin Oral Implants Res. 2016 Oct;27(10):1274-1282. doi: 10.1111/clr.12732. Epub 2015 Nov 23. PMID 26592859
- [Result] Weltman NJ, Al-Attar Y, Cheung J, Duncan DP, Katchky A, Azarpazhooh A, Abrahamyan L. MANAGEMENT OF DENTAL EXTRACTIONS IN PATIENTS TAKING WARFARIN AS ANTICOAGULANT TREATMENT: A SYSTEMATIC REVIEW. J Can Dent Assoc. 2015;81:f20. PMID 26679334
- [Result] Cai J, Ribkoff J, Olson S, Raghunathan V, Al-Samkari H, DeLoughery TG, Shatzel JJ. The many roles of tranexamic acid: An overview of the clinical indications for TXA in medical and surgical patients. Eur J Haematol. 2020 Feb;104(2):79-87. doi: 10.1111/ejh.13348. Epub 2019 Dec 16. PMID 31729076
- [Result] Ker K, Beecher D, Roberts I. Topical application of tranexamic acid for the reduction of bleeding. Cochrane Database Syst Rev. 2013 Jul 23;2013(7):CD010562. doi: 10.1002/14651858.CD010562.pub2. PMID 23881695
- [Result] Cankaya D, Dasar U, Satilmis AB, Basaran SH, Akkaya M, Bozkurt M. The combined use of oral and topical tranexamic acid is a safe, efficient and low-cost method in reducing blood loss and transfusion rates in total knee arthroplasty. J Orthop Surg (Hong Kong). 2017 Jan;25(1):2309499016684725. doi: 10.1177/2309499016684725. PMID 28176599
- [Result] Perdigao JP, de Almeida PC, Rocha TD, Mota MR, Soares EC, Alves AP, Sousa FB. Postoperative bleeding after dental extraction in liver pretransplant patients. J Oral Maxillofac Surg. 2012 Mar;70(3):e177-84. doi: 10.1016/j.joms.2011.10.033. PMID 22374059
- [Result] Ockerman A, Vanhaverbeke M, Miclotte I, Belmans A, Vanassche T, Politis C, Jacobs R, Verhamme P. Tranexamic acid to reduce bleeding after dental extraction in patients treated with non-vitamin K oral anticoagulants: design and rationale of the EXTRACT-NOAC trial. Br J Oral Maxillofac Surg. 2019 Dec;57(10):1107-1112. doi: 10.1016/j.bjoms.2019.10.297. Epub 2019 Oct 25. PMID 31669068
- [Result] Patatanian E, Fugate SE. Hemostatic mouthwashes in anticoagulated patients undergoing dental extraction. Ann Pharmacother. 2006 Dec;40(12):2205-10. doi: 10.1345/aph.1H295. Epub 2006 Nov 7. PMID 17090725
- [Result] Couto EV, Ballin CR, Sampaio CP, Maeda CA, Ballin CH, Dassi CS, Miura LY. Experimental study on the effects of bismuth subgallate on the inflammatory process and angiogenesis of the oral mucosa. Braz J Otorhinolaryngol. 2016 Jan-Feb;82(1):17-25. doi: 10.1016/j.bjorl.2014.12.009. Epub 2015 Oct 27. PMID 26614041
- [Result] Thorisdottir H, Ratnoff OD, Maniglia AJ. Activation of Hageman factor (factor XII) by bismuth subgallate, a hemostatic agent. J Lab Clin Med. 1988 Oct;112(4):481-6. PMID 3171356
- [Result] Maniglia AJ, Kushner H, Cozzi L. Adenotonsillectomy. A safe outpatient procedure. Arch Otolaryngol Head Neck Surg. 1989 Jan;115(1):92-4. doi: 10.1001/archotol.1989.01860250094034. PMID 2909235
- [Result] Radoi L, Hajage D, Giboin C, Maman L, Monnet-Corti V, Descroix V, Mahe I. Perioperative management of oral anticoagulated patients undergoing an oral, implant, or periodontal procedure: a survey of practices of members of two dental scientific societies, the PRADICO study. Clin Oral Investig. 2019 Dec;23(12):4311-4323. doi: 10.1007/s00784-019-02877-1. Epub 2019 Mar 19. PMID 30887189
- [Result] Bacci C, Berengo M, Favero L, Zanon E. Safety of dental implant surgery in patients undergoing anticoagulation therapy: a prospective case-control study. Clin Oral Implants Res. 2011 Feb;22(2):151-6. doi: 10.1111/j.1600-0501.2010.01963.x. Epub 2010 Oct 13. PMID 20946205
- [Result] Wilson W, Taubert KA, Gewitz M, Lockhart PB, Baddour LM, Levison M, Bolger A, Cabell CH, Takahashi M, Baltimore RS, Newburger JW, Strom BL, Tani LY, Gerber M, Bonow RO, Pallasch T, Shulman ST, Rowley AH, Burns JC, Ferrieri P, Gardner T, Goff D, Durack DT; American Heart Association Rheumatic Fever, Endocarditis, and Kawasaki Disease Committee; American Heart Association Council on Cardiovascular Disease in the Young; American Heart Association Council on Clinical Cardiology; American Heart Association Council on Cardiovascular Surgery and Anesthesia; Quality of Care and Outcomes Research Interdisciplinary Working Group. Prevention of infective endocarditis: guidelines from the American Heart Association: a guideline from the American Heart Association Rheumatic Fever, Endocarditis, and Kawasaki Disease Committee, Council on Cardiovascular Disease in the Young, and the Council on Clinical Cardiology, Council on Cardiovascular Surgery and Anesthesia, and the Quality of Care and Outcomes Research Interdisciplinary Working Group. Circulation. 2007 Oct 9;116(15):1736-54. doi: 10.1161/CIRCULATIONAHA.106.183095. Epub 2007 Apr 19. PMID 17446442
- [Result] Sannino G, Cappare P, Montemezzi P, Alfieri O, Pantaleo G, Gherlone E. Postoperative bleeding in patients taking oral anticoagulation therapy after 'All-on-four' rehabilitation: A case-control study. Int J Oral Implantol (Berl). 2020;13(1):77-87. PMID 32186289
- [Result] Guyatt GH, Akl EA, Crowther M, Gutterman DD, Schuunemann HJ; American College of Chest Physicians Antithrombotic Therapy and Prevention of Thrombosis Panel. Executive summary: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):7S-47S. doi: 10.1378/chest.1412S3. No abstract available. PMID 22315257
- [Result] Zanon E, Martinelli F, Bacci C, Cordioli G, Girolami A. Safety of dental extraction among consecutive patients on oral anticoagulant treatment managed using a specific dental management protocol. Blood Coagul Fibrinolysis. 2003 Jan;14(1):27-30. doi: 10.1097/00001721-200301000-00006. PMID 12544725
- [Result] Broekema FI, van Minnen B, Jansma J, Bos RR. Risk of bleeding after dentoalveolar surgery in patients taking anticoagulants. Br J Oral Maxillofac Surg. 2014 Mar;52(3):e15-9. doi: 10.1016/j.bjoms.2014.01.006. Epub 2014 Jan 30. PMID 24485810
- [Result] Di Minno A, Frigerio B, Spadarella G, Ravani A, Sansaro D, Amato M, Kitzmiller JP, Pepi M, Tremoli E, Baldassarre D. Old and new oral anticoagulants: Food, herbal medicines and drug interactions. Blood Rev. 2017 Jul;31(4):193-203. doi: 10.1016/j.blre.2017.02.001. Epub 2017 Feb 5. PMID 28196633
- [Result] Schmitt CM, Rusche B, Clemm R, Neukam FW, Buchbender M. Management of anticoagulated patients in dentoalveolar surgery: a clinical comparative study. Clin Oral Investig. 2020 Aug;24(8):2653-2662. doi: 10.1007/s00784-019-03124-3. Epub 2019 Nov 12. PMID 31713746
- [Result] Soares EC, Costa FW, Bezerra TP, Nogueira CB, de Barros Silva PG, Batista SH, Sousa FB, Sa Roriz Fonteles C. Postoperative hemostatic efficacy of gauze soaked in tranexamic acid, fibrin sponge, and dry gauze compression following dental extractions in anticoagulated patients with cardiovascular disease: a prospective, randomized study. Oral Maxillofac Surg. 2015 Jun;19(2):209-16. doi: 10.1007/s10006-014-0479-9. Epub 2014 Dec 21. PMID 25528251
- [Result] Ferrieri GB, Castiglioni S, Carmagnola D, Cargnel M, Strohmenger L, Abati S. Oral surgery in patients on anticoagulant treatment without therapy interruption. J Oral Maxillofac Surg. 2007 Jun;65(6):1149-54. doi: 10.1016/j.joms.2006.11.015. PMID 17517299
- [Result] Kim SH, Tramontina VA, Papalexiou V, Luczyszyn SM. Bismuth subgallate as a topical hemostatic agent at palatal donor sites. Quintessence Int. 2010 Sep;41(8):645-649. PMID 20657853
- [Result] Callanan V, Curran AJ, Smyth DA, Gormley PK. The influence of bismuth subgallate and adrenaline paste upon operating time and operative blood loss in tonsillectomy. J Laryngol Otol. 1995 Mar;109(3):206-8. doi: 10.1017/s0022215100129706. PMID 7745335
- [Result] Scully C, Hobkirk J, Dios PD. Dental endosseous implants in the medically compromised patient. J Oral Rehabil. 2007 Aug;34(8):590-9. doi: 10.1111/j.1365-2842.2007.01755.x. PMID 17650169
- [Result] Diz P, Scully C, Sanz M. Dental implants in the medically compromised patient. J Dent. 2013 Mar;41(3):195-206. doi: 10.1016/j.jdent.2012.12.008. Epub 2013 Jan 11. PMID 23313715
- [Result] Proietti R, Porto I, Levi M, Leo A, Russo V, Kalfon E, Biondi-Zoccai G, Roux JF, Birnie DH, Essebag V. Risk of pocket hematoma in patients on chronic anticoagulation with warfarin undergoing electrophysiological device implantation: a comparison of different peri-operative management strategies. Eur Rev Med Pharmacol Sci. 2015 Apr;19(8):1461-79. PMID 25967723
- [Result] Bajkin BV, Urosevic IM, Stankov KM, Petrovic BB, Bajkin IA. Dental extractions and risk of bleeding in patients taking single and dual antiplatelet treatment. Br J Oral Maxillofac Surg. 2015 Jan;53(1):39-43. doi: 10.1016/j.bjoms.2014.09.009. Epub 2014 Oct 11. PMID 25311541
- [Result] DeClerck D, Vinckier F, Vermylen J. Influence of anticoagulation on blood loss following dental extractions. J Dent Res. 1992 Feb;71(2):387-90. doi: 10.1177/00220345920710020701. PMID 1532608
- [Result] Dunn AS, Turpie AG. Perioperative management of patients receiving oral anticoagulants: a systematic review. Arch Intern Med. 2003 Apr 28;163(8):901-8. doi: 10.1001/archinte.163.8.901. PMID 12719198